CLINICAL TRIAL: NCT00691860
Title: Randomized, Controlled, Prospective Study of the Use of a Mesh to Prevent Parastomal Hernia
Brief Title: Use of a Mesh to Prevent Parastomal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Xavier Serra-Aracil, Corporacio Sanitaria Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSPT-SerraA-01
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2008-06

CONDITIONS: Parastomal Hernia
Keywords: Parastomal hernias; Tolerance of lightweight meshes; Paracolostomy hernias; Peristomal hernias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients receiving conventional sigmoid end colostomy plus a lightweight mesh Ultrapro®
  Interventions: Device: Mesh (Ultrapro ®); Procedure: Conventional sigmoid end colostomy
- 2 (Other): Patients receiving conventional sigmoid end colostomy, without mesh
  Interventions: Procedure: Conventional sigmoid end colostomy

INTERVENTIONS:
Device: Mesh (Ultrapro ®) — In the mesh group, the mesh was placed in the sublay position, above the peritoneum and the posterior rectus sheath of the rectus abdominis muscles, with a minimum of 5 cm of mesh around the colostomy
  Other Names: Ultrapro ®
  Arms: 1
Procedure: Conventional sigmoid end colostomy — Patients receiving conventional sigmoid end colostomy, without mesh

SUMMARY:
Randomized, controlled, prospective study of 54 patients receiving surgery for cancer of the lower third of the rectum with a permanent end colostomy. The aim of the study was to reduce parastomal hernia (PH) occurrence by implanting a lightweight mesh in the sublay position. Patients were followed up a) clinically and b) radiologically by means of abdominal CT. In the clinical follow-up, hernias were observed in four out of 27 patients (14.8%) in the study group and in eleven out of 27 (40.7%) in the control group (p=0.03). The implantation of the mesh reduces the appearance of PH, is well tolerated, and does not increase morbidity

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for permanent end colostomy to treat cancer of the lower third of the rectum,
* Aged over 18,
* Charlson comorbidity index below 7
* Elective surgery
* Radical surgery

Exclusion Criteria:

* Loop colostomies,
* Emergency surgery,
* Body mass index above 35 kg/sq.m.,
* Palliative surgery,
* Hepatic cirrhosis,
* Severe COPD (requiring home oxygen treatment),
* Corticoid treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-04; Primary Completion 2007-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
the reduction in the incidence of Parastomal Hernia after the mesh placement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Navarro-Soto, MD, Study Chair — Corporacio Sanitaria Parc Tauli